CLINICAL TRIAL: NCT02234232
Title: Exercise in the Dialysis Unit: a Randomized Factorial Pilot Study on the Feasibility and Safety of Intradialytic Exercise
Brief Title: The Feasibility and Safety of an Intradialytic Exercise Program: DIALY-SIZE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Alberta Innovates Health Solutions (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Other
Other Study IDs: RES0016810; RES0018218 (Other Grant/Funding Number: Alberta Innovates Health Solutions)
Record Dates: First submitted 2014-09-02; First posted 2014-09-09 (Estimated); Last update posted 2022-07-19 (Actual); Status verified 2015-04

CONDITIONS: End-stage Renal Disease
Keywords: Hemodialysis; Exercise, aerobic; Exercise, resistance; Intradialytic; Randomized Controlled Trial; Safety; Quality of life; Physical performance
MeSH Terms: conditions — Kidney Failure, Chronic; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Aerobic exercise (Experimental): Cycling-participants will exercise for 15 minutes at the initial session followed by a weekly increase of 2 min and 3 seconds over 12 weeks. Participants will exercise 3 times per week and an intensity of "somewhat hard" (12-14 on the Borg scale). All exercises will be performed during hemodialysis.
  Interventions: Behavioral: Exercise
- Resistance (Experimental): Resistance training of lower limbs using ankle weights. Participants will complete 10-15 repetitions of 4 lower limb exercises: knee extension, straight leg raise, hip abduction, and hip flexion. Exercises will progress from 1 set of each exercise up to 3 sets of each exercise and with weight. Participants will exercise 3 times per week and an intensity of "somewhat hard" (12-14 on the Borg scale). All exercises will be performed during hemodialysis.
  Interventions: Behavioral: Exercise
- Combined aerobic and resistance (Experimental): Participants will complete both the aerobic (cycling) and resistance (ankle weights) exercise prescriptions.
  Interventions: Behavioral: Exercise
- Flexibility (Active Comparator): A non-progressive flexibility regimen using a stretch band. Participants will perform 2 sets of the following exercises: seated pelvic tilt, seated calf stretch, supine hamstring stretch, and supine gluteal stretch. Participants will exercise 3 times per week and an intensity of "very light" (9 on the Borg scale). All exercises will be performed during hemodialysis.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Each exercise will be performed during the first 2.5 hours of the participant's hemodialysis session. Exercises are semi supervised: the kinesiologist will supervise the initial three exercise sessions, any session that requires a change to the exercise prescription and on a minimum of a weekly basis.
  Other Names: Monark ergometers; TherapyTrainer ergometers; TheraBand Stretch Strap; The Cuff ankle weights

SUMMARY:
The primary aim of this pilot study is to evaluate the feasibility and safety of four different types of intradialytic exercise (exercise performed during dialysis) programs: resistance, aerobic, combined resistance and aerobic, and flexibility (attention control). The secondary aim of the study is to estimate the effect of aerobic and resistance exercise, each compared with the attention control on: health-related quality of life, tests of physical performance, strength, and physical activity outside of the dialysis unit. The results of this study will be used to inform the planning of a full-scale efficacy study.

DETAILED DESCRIPTION:
Recruitment: participants will be recruited by a study coordinator during their regular hemodialysis shift. This is a quaternary outpatient dialysis unit serving approximately 110 patients.

Randomization and allocation: we will use a permuted block design with randomly varied block sizes of eight and twelve. The randomization sequence will be computer generated and randomization to one of the 4 groups will be on a 1:1:1:1 ratio. Allocation is concealed in serially numbered, opaque, sealed envelopes.

Data collection: demographic data, length of time of hemodialysis, cause of ESRD, access type, comorbidities, number of medications, functional status, comorbidities, and dialysis prescription will be collected. The laboratory values and dialysis prescription will be collected from the dialysis unit chart using the most recent monthly blood-work and from the provincial laboratory repository. The amount and intensity of exercise that was performed as well as the participant's heart rate and blood pressure during the exercise session will be recorded at each exercise session. The exercise forms from each participant's dialysis session will be reviewed weekly for missing data. Forms with any empty field will be classified as incomplete and where possible, the appropriate staff will be asked to verify the query.

The occurrence of adverse events will be collected from all four randomization groups.The hemodialysis run-sheet, nursing notes, and exercise data collection form will be reviewed weekly for the occurence of adverse events. Hemodialysis unit staff and the exercise trainer have been instructed to report adverse events (defined a priori) as they occur. In addition, prior to each exercise session, participants will be asked if they have had any new health problems or symptoms since their last exercise session.

Missing data: conditional on the participant's consent, outcome data will be collected from all participants who drop out. For those participants who do not wish to be followed or who have missing data, baseline data will be carried forward.

Safety: due to the short duration and small size of this study, a formal safety and trial management board will not be established. A nephrologist who is not affiliated with the study will review all SAEs as they occur. The nephrologist will then determine if the SAE was associated with the intervention and whether the individual's participation requires modification or discontinuation.

Statistical analysis plan: descriptive statistics will be used to compare the clinical characteristics of the four groups at baseline. All analyses will follow the intention to treat principle.

Safety: in a primary analysis, adverse events will be reported as the number of events directly related to the intervention compared to control, by randomization group. In a secondary analysis, all adverse events that occurred during the study will be analyzed. The frequency of events will be compared using ANOVA or Kruskal-Wallis where appropriate, and with appropriate post-hoc tests to detect differences between randomization groups.

To explore the effect of aerobic and resistance exercise on components of HRQOL we will estimate the absolute change in score at 12 weeks relative to baseline in the physical component summary score (PCS), the mental component summary score (MCS), and the kidney-disease specific score (KDCS). We will report the absolute change in sub-scores for each of the component summary scores. We will use the same method to estimate the difference in scores on the tests of physical performance and strength. Assuming there is no statistical interaction (no indication in the literature), we will estimate the efficacy of the aerobic intervention by comparing all participants who received aerobic exercise with all groups that did not (aerobic and combined exercise groups versus resistance and control exercise groups) and similarly for the resistance-training group. Final scores will be compared using analysis of covariance (ANCOVA) adjusting for the baseline scores and both main effect terms. The final score will be presented as the adjusted difference in the means. To correct for multiple comparisons in the combined exercise group, based on the Bonferroni procedure a significance level of less than 0.025 will be considered significant. The same method will be used to analyze differences in the tests of physical functioning and strength. The interaction will be estimated in a secondary analysis. Due to the small sample size, no subgroup analysis will be performed.

ELIGIBILITY:
Inclusion Criteria:

* adult (age ≥18)
* dialysis dependent for ≥ 3 consecutive months
* receiving ≥ 3 dialysis treatments per week
* mobile (any distance and can be with the assistance of an aid)
* at least one non-prosthetic and functional limb
* stable during hemodialysis treatment (assessed by hemodialysis unit staff and the study physician)
* capable of providing consent

Exclusion Criteria:

* currently enrolled in a clinical trial
* missing an average of more than 2 shifts per month
* planned move or modality change within the next 4 months
* currently enrolled in a structured exercise program
* scheduled hospitalization for > 1 week
* any uncontrolled medical condition that would preclude participation in a low/moderate intensity exercise program (e.g. unstable angina, uncontrolled hypertension, severe valvular heart disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2014-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
The number of participants with an adverse event | Change from baseline to 12 weeks
  among each of the intervention groups, the number of participants with and type of adverse events will be compared to control. Adverse events are defined a priori and classified as either i. Serious adverse events (cardiac event e.g. arrhythmia, myocardial infarction; death; hospitalization; disability; any life threatening event) or ii. Adverse events (musculoskeletal injury; hypoglycemia; hypotension, defined as a decrease in systolic blood pressure by ≥20 mm Hg with symptoms or requiring an intervention during exercise; hypertension, define as a sustained elevation in blood pressure of >200 mmHg systolic or >110 diastolic; dialysis access complications (e.g. re-needling, hematosis, thrombosis); and any staff intervention beyond minimum ultrafiltration.
Adherence to the exercise protocol | At 12 weeks
  To indicate the willingness of participants to engage in intradialytic exercise, adherence will be reported as the proportion of exercise sessions that were initiated out of the total number of sessions prescribed (defined as ≥ 70% of exercise sessions). To measure the amount of exercise that was actually performed, adherence will be defined as the number of sessions that were completed out of the total number of sessions prescribed (defined as ≥ 70% of exercise sessions). Adherence will be reported according to randomization groups.
The number of dropouts | At the end of the study, 6 months
  A dropout is defined as a participant who leaves the study for any reason prior to completing the 12-week (36 session) exercise program. All reasons for drop out will be reported.
Human activity profile | Change from baseline to 12 weeks
  To evaluate if an exercise program would influence the level of daily physical activity in this population, the difference in the amount of daily physical activity performed outside of the HD unit at baseline and at 12 weeks will be measured.
The number of participants who adopted the other group's exercise | Change from baseline and 12 weeks
  Due the open nature of the dialysis unit, participants are aware of other participant's exercise assignments. To measure the effect of contamination, we will obtain this information from participants at the end of the study through an anonymized questionnaire.
The proportion of patients that would continue their current intradialytic exercise program after the study is over. | At the end of the study, 6 months.
  Defined as ≥50% of participants reporting that they would like to continue their current intradialytic exercise program after the study is over. This information will be collected at the end of the study using an anonymized questionnaire

SECONDARY OUTCOMES:
Health-related quality of life | Change from baseline to 12 weeks
  Using the KDQOL SF-36, the change in the summary and component scores.
Physical performance | Change from baseline to 12 weeks
  The Short Physical Performance Battery
The six minute walk test | Change from baseline to 12 weeks
Number of chair stands completed in 30 seconds | Change from baseline to 12 weeks
Strength, one repetition maximum | Change from baseline to 12 weeks

OTHER OUTCOMES:
Physical performance | Pre/post (12 weeks)
  Strength (1 repetition maximum)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Thompson, MD, Principal Investigator — University of Alberta; Scott Klarenbach, MD, Principal Investigator — University of Alberta; Marcello Tonelli, MD, Principal Investigator — University of Calgary
Locations (1):
- University of Alberta Hospital, outpatient dialysis unit, Edmonton, Alberta, Canada

REFERENCES:
- [Result] Thompson S, Klarenbach S, Molzahn A, Lloyd A, Gabrys I, Haykowsky M, Tonelli M. Randomised factorial mixed method pilot study of aerobic and resistance exercise in haemodialysis patients: DIALY-SIZE! BMJ Open. 2016 Sep 6;6(9):e012085. doi: 10.1136/bmjopen-2016-012085. PMID 27601500
- [Derived] Bernier-Jean A, Beruni NA, Bondonno NP, Williams G, Teixeira-Pinto A, Craig JC, Wong G. Exercise training for adults undergoing maintenance dialysis. Cochrane Database Syst Rev. 2022 Jan 12;1(1):CD014653. doi: 10.1002/14651858.CD014653. PMID 35018639